CLINICAL TRIAL: NCT02126956
Title: Single-center, Open-label Study With 14C-labeled ACT-128800 to Investigate the Mass Balance, Pharmacokinetics, and Metabolism Following Single Oral Administration to Healthy Male Subjects
Brief Title: Mass Balance, Pharmacokinetics, and Metabolism of 14C-labeled ACT-128800 Administered to Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AC-058-106
Record Dates: First submitted 2014-04-29; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Pharmacokinetics
Keywords: ACT-128800
MeSH Terms: interventions — ponesimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACT-128800 (Experimental): Subjects received a single oral dose of 40 mg 14C-labeled ACT-128800 (one capsule)
  Interventions: Drug: ACT-128800

INTERVENTIONS:
Drug: ACT-128800 — ACT-128800 was supplied as a powder mix in hard gelatin capsules for oral administration. The capsules contained a co-precipitated mixture of non-radiolabeled and 14C-labeled ACT-128800 formulated at a dose strength of 40 mg with a maximum radioactive content of 102 μCi (3.79 MBq).

SUMMARY:
The study was conducted to investigate the metabolism and mass balance of ACT-128800, and to identify the elimination pathways (metabolism and excretion) of ACT-128800 and compare them with the known metabolic profiles of ACT-128800 in animals.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Male and aged between 45 and 65 years (inclusive) at screening.
* No clinically significant findings on physical examination performed at screening.
* Body mass index (BMI) between 18-28 kg/m^2 (inclusive) at screening.
* Systolic blood pressure 100-145 mmHg, diastolic blood pressure 50-90 mmHg, and heart rate 55-90 bpm (inclusive), measured on the leading arm, after 5 minutes in the supine position at screening. These criteria should also be met before the administration of the first dose.
* 12-lead electrocardiogram without clinically relevant abnormalities at screening.
* Clinical chemistry, hematology, and urinalysis results not deviating from the normal range to a clinically relevant extent at screening.
* Negative results from urine drug screen at screening.
* Ability to communicate well with the investigator in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Known hypersensitivity to any excipients of the drug formulation.
* Treatment with another investigational drug within the 3 months prior to screening.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* Excessive caffeine consumption, defined as ≥ 800 mg per day at screening.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drug.
* Smoking within the 3 months prior to screening.
* Any immunosuppressive treatment within 6 weeks before study drug administration.
* Previous treatment with any prescribed or over-the-counter medications (including herbal medicines such as St John's Wort) within 2 weeks prior to screening.
* Loss of 250 mL or more of blood within the 3 months prior to screening.
* Lymphopenia (< 1,100 lymphocytes/μL).
* Viral, fungal, bacterial or protozoal infection within 4 weeks before study drug administration.
* Positive hepatitis B or hepatitis C serology, except for vaccinated subjects, at screening.
* Positive human immunodeficiency virus serology at screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Legal incapacity or limited legal capacity at screening.
* Exposure to artificial ionizing radiation (e.g., X-ray, thyroid scan, study with radiolabeled compound) in the 12-month period before screening.
* A history of clinically relevant constipation (defined as lasting more than 3 days) in the 4-week period before screening.

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Cumulative recovery of total radioactivity expressed as a percentage of the administered dose (mass balance) in the urine | Up to end of study, approximately 240 hours
  On Day 1, immediately prior to the intake of study drug, subjects were instructed to empty their bladders. Thereafter, following drug intake all urine produced was collected for 10 days up to Day 11 (morning). Following administration of 14C-ACT-128800, urine samples were collected in three consecutive 8-hour intervals, from 0-8 h, 8-16 h, and 16-24 h. From Day 2 to Day 10 (inclusive), urine samples were collected at 24-hour intervals. In case of an extended observation period, urine samples were also collected at 24-hour intervals. The total amount of radioactivity was measured using a liquid scintillation counter.
Cumulative recovery of total radioactivity expressed as a percentage of the administered dose (mass balance) in the faeces | Up to end of study, approximately 240 hours
  Between Day -3 and Day -1, a baseline faeces sample was collected in a light-protected polypropylene box from each subject.
  From Day 1 (post-dose) to Day 10 (inclusive), all faeces samples and the toilet paper were collected in pre-weighed, light-protected polypropylene boxes. Each faeces sample was collected in a separate box and weighed. The weight of the sample and the time of collection were recorded. All faecal samples were frozen as soon as possible and stored in an upright position at -70 °C or below.The total amount of radioactivity was measured using a liquid scintillation counter.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of 14C-radioactivity in whole blood | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.0 mL was used for measurement of radioactivity. The amount of radioactivity was measured using a liquid scintillation counter. The measured radioactivity was used to directly obtain Cmax.
Time to maximum concentration (tmax) of 14C-radioactivity in whole blood | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.0 mL was used for measurement of radioactivity. The amount of radioactivity was measured using a liquid scintillation counter. The measured radioactivity was used to directly obtain tmax.
Area under the plasma concentration-time curve (AUC(0-t)) of 14C-radioactivity in whole blood | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.0 mL was used for measurement of radioactivity. The amount of radioactivity was measured using a liquid scintillation counter. AUC(0-t) was calculated according to the linear trapezoidal rule, using the measured concentration-time values above the limit of quantification.
Area under the plasma concentration-time curve (AUC(0-infinity)) of 14C-radioactivity in whole blood | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.0 mL was used for measurement of radioactivity. The amount of radioactivity was measured using a liquid scintillation counter. AUC(0-infinity) was calculated by combining AUC(0-t) and AUC(extra). AUC(extra) represents an extrapolated value obtained by Ct/λz,, where Ct is the last concentration above the limit of quantification and λz, represents the terminal elimination rate constant determined by log-linear regression analysis of the measured concentrations in the terminal elimination phase.
Half life (t1/2) of 14C-radioactivity in whole blood | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.0 mL was used for measurement of radioactivity. The amount of radioactivity was measured using a liquid scintillation counter. t1/2 was calculated as follows: t1/2 = ln 2/λz, where ln 2 is the natural log of 2 (approximately 0.693).
Maximum concentration (Cmax) of 14C-radioactivity in plasma | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.0 mL was used for measurement of radioactivity. The amount of radioactivity was measured using a liquid scintillation counter. The measured radioactivity was used to directly obtain Cmax.
Time to maximum concentration (tmax) of 14C-radioactivity in plasma | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.0 mL was used for measurement of radioactivity. The amount of radioactivity was measured using a liquid scintillation counter. The measured radioactivity was used to directly obtain tmax.
Area under the plasma concentration-time curve (AUC(0-t)) of 14C-radioactivity in plasma | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.0 mL was used for measurement of radioactivity. The amount of radioactivity was measured using a liquid scintillation counter. AUC(0-t) was calculated according to the linear trapezoidal rule, using the measured concentration-time values above the limit of quantification.
Area under the plasma concentration-time curve (AUC(0-infinity)) of 14C-radioactivity in plasma | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.0 mL was used for measurement of radioactivity. The amount of radioactivity was measured using a liquid scintillation counter. AUC(0-infinity) was calculated by combining AUC(0-t) and AUC(extra). AUC(extra) represents an extrapolated value obtained by Ct/λz,, where Ct is the last concentration above the limit of quantification and λz, represents the terminal elimination rate constant determined by log-linear regression analysis of the measured concentrations in the terminal elimination phase.
Half life (t1/2) of 14C-radioactivity in plasma | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.0 mL was used for measurement of radioactivity.The amount of radioactivity was measured using a liquid scintillation counter. t1/2 was calculated as follows: t1/2 = ln 2/λz, where ln 2 is the natural log of 2 (approximately 0.693).
Maximum concentration (Cmax) of ACT-12880 in plasma | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.7 mL was used for measurement of ACT-12880 concentration. The concentration of ACT-128800 was determined using a validated liquid chromatography-tandem mass spectrometry assay was used to directly obtain Cmax.
Time to maximum concentration (tmax) of ACT-12880 in plasma | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.7 mL was used for measurement of ACT-12880 concentration. The concentration of ACT-128800 was determined using a validated liquid chromatography-tandem mass spectrometry assay was used to directly obtain tmax.
Area under the plasma concentration-time curve (AUC(0-t)) of ACT-12880 in plasma | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.7 mL was used for measurement of ACT-12880 concentration. The concentration of ACT-128800 was determined using a validated liquid chromatography-tandem mass spectrometry assay . AUC(0-t) was calculated according to the linear trapezoidal rule, using the measured concentration-time values above the limit of quantification.
Area under the plasma concentration-time curve (AUC(0-infinity)) of ACT-12880 in plasma | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.7 mL was used for measurement of ACT-12880 concentration. The concentration of ACT-128800 was determined using a validated liquid chromatography-tandem mass spectrometry assay . AUC(0-infinity) was calculated by combining AUC(0-t) and AUC(extra). AUC(extra) represents an extrapolated value obtained by Ct/λz,, where Ct is the last concentration above the limit of quantification and λz, represents the terminal elimination rate constant determined by log-linear regression analysis of the measured concentrations in the terminal elimination phase.
Half life (t1/2) of ACT-12880 in plasma | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.7 mL was used for measurement of ACT-12880 concentration. The concentration of ACT-128800 was determined using a validated liquid chromatography-tandem mass spectrometry assay . t1/2 was calculated as follows: t1/2 = ln 2/λz, where ln 2 is the natural log of 2 (approximately 0.693).
Total lymphocyte count | Up to end of study, approximately 240 hours
  Blood samples were collected from an antecubital vein by direct venipuncture or via an intravenous catheter at various time points up to the end of study. An aliquot of 2.7 mL was used for measurement of lymphocyte count
Change in systolic blood pressure from baseline up to end of study | Up to end of study, approximately 240 hours
  Blood pressure was measured at various time points up to the end of study using an automatic oscillometric device. Measurements were taken with the subject in the supine position after a resting period of at least 5 minutes. The leading (writing) arm was used for all blood pressure measurements.
Change in diastolic blood pressure from baseline up to end of study | Up to end of study, approximately 240 hours
  Blood pressure was measured at various time points up to the end of study using an automatic oscillometric device. Measurements were taken with the subject in the supine position after a resting period of at least 5 minutes. The leading (writing) arm was used for all blood pressure measurements.
Change in heart rate from baseline up to end of study | Up to end of study, approximately 240 hours
  Heart rate was measured at various time points up to the end of study using an automatic oscillometric device. Measurements were taken with the subject in the supine position after a resting period of at least 5 minutes. The leading (writing) arm was used for all blood pressure measurements.
Change in body temperature from baseline up to end of study | Up to end of study, approximately 240 hours
  Body temperature was measured at various time points up to the end of study.
Change in body weight from baseline to end of study | Up to end of study, approximately 240 hours
  Body weight was measured at baseline and at end of study using the same weighing scales for all subjects. The weighing scales had a precision of at least 0.5 kg.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Brossard, PhD, Study Director — Actelion
Locations (1):
- Swiss Pharma Contract, Allschwil, Switzerland